CLINICAL TRIAL: NCT01657383
Title: Surgical Outcomes Database for Faculty of Hepatopancreatico Biliary Surgery
Brief Title: Surgical Outcomes Database For Faculty of Hepatopancreatic Biliary Surgery
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 04-12-02E
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2017-07

CONDITIONS: Cancer of Liver; Pancreatic Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hepatopancreaticobiliary (HPB) Surgery Patients: Patients undergoing surgical HPB procedures
  Interventions: Procedure: HPB Surgery

INTERVENTIONS:
Procedure: HPB Surgery — Hepatopancreatico Biliary Surgery

SUMMARY:
The collection of data regarding patient outcomes after surgical intervention creates imperative knowledge to include surgeon performance, cost analysis, base for surgical research and publication, which in turn assist surgeons to improve the standard of care utilizing evidence-based practice.

DETAILED DESCRIPTION:
The concept of disease management stems from a logical evolution in the field of outcomes applications by healthcare provides is the concept of disease management. The basic premise of disease management is that there is a more optimal way to manage patients in order to reduce costs and improve health outcomes. The data collected from patient-reported outcomes allows the physician and staff to screen for specific health conditions, monitor patients individually, evaluate outcomes for specific groups, assess quality of care, determine impact of intervention and predict outcomes. Most of the follow-up results from this study will be obtained directly from the patient during follow-up visits, but other information may be obtained from medical records.

Evaluation of the surgical database Application will identify both patient and procedural variables that can predict adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are Hepatopancreatico Biliary surgical patients.

Exclusion Criteria:

* Patients that are not Hepatopancreatico Biliary surgical patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatopancreatico Biliary surgical patients.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Surgical Outcome | 1 year
  Quality of life evaluation after surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David A Iannitti, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Health System, Charlotte, North Carolina, United States